CLINICAL TRIAL: NCT02703233
Title: A Randomized Control Trial of Nitrous Oxide Use in the Emergency Department
Brief Title: Effectiveness of Nitrous Oxide in the ED
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Feasibility
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 602966
Record Dates: First submitted 2016-02-24; First posted 2016-03-09 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Lacerations; Abscess
MeSH Terms: conditions — Lacerations; Abscess | interventions — Nitrous Oxide; Oxygen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrous Oxide (Active Comparator): Patients receive nitrous oxide via mask.
  Interventions: Drug: Nitrous Oxide
- Placebo (Oxygen) (Placebo Comparator): Patients receive oxygen via mask.
  Interventions: Other: Oxygen

INTERVENTIONS:
Drug: Nitrous Oxide
  Arms: Nitrous Oxide
Other: Oxygen
  Arms: Placebo (Oxygen)

SUMMARY:
This will be a randomized control trial. All patients for whom an emergency provider determines that abscess drainage or laceration repair are necessary will be considered for enrollment. The provider must be willing to participate in the study and be certified to use Nitrous oxide. The investigators providers completed a training course to be certified to use Nitrous oxide. The patient must be age 18 or greater, consent to participate in the study, and be able to complete a satisfaction survey. If the patient states there is a possibility of pregnancy, the investigators will regress to our standard of care and perform a urine pregnancy test. Patients with a first trimester pregnancy will be excluded. Patients who agree to enroll in the study will be randomized to Nitrous oxide versus oxygen (to be administered through the same system), and will complete a survey after the procedure, as will the provider. There will be a separate block randomization for each procedure. Providers may select other agents of choice for analgesia/sedation, such as local anesthesia, and pain medications, based on their clinical judgment. If the patient appears to have inadequate analgesia during the procedure, the provider can elect to treat as is typically done (pain medications or local anesthetics) at their discretion. The survey will ask patients to give a self-reported pain score before and during their procedure (both to be completed after the procedure). It will also ask the patient/guardian and provider for a satisfaction level with the analgesia during the procedure. In addition, side effects and procedure start and stop time will also be documented. In addition to the survey, the investigators will document clinical characteristics including diagnosis, size of laceration or abscess, additional medications required and dosages, comorbidities, age, and gender. Other data that will be gathered will include which adjunctive analgesics/anesthetics were used.

ELIGIBILITY:
Inclusion Criteria:

Patients with:

* A laceration or an abscess requiring primary repair or incision and drainage respectively, per the treating provider

Exclusion Criteria:

* Age < 18 years
* First trimester pregnancy
* Inability to obtain written informed consent from subject or surrogate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-03 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Pain Assessment Scale (0-10) | 0-20 minutes after drug administration
  Pain score will be collected after drug administration

SECONDARY OUTCOMES:
Provider satisfaction score | 0-20 minutes after drug administration
  Provider satisfaction collected via survey post drug administration
Patient satisfaction | 0-20 minutes after drug administration
  Patient satisfaction collected via survey post drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Brian Levine, MD, Principal Investigator — Christiana Care Health Services

IPD SHARING:
Plan to Share IPD: No